CLINICAL TRIAL: NCT00852176
Title: Best Vascular P000018 Post-approval Study: Retrospective Long-term Safety and Efficacy Study of the Beta-Cath(TM) 3.5F System
Brief Title: Retrospective Long-term Safety and Efficacy Study of the Beta-Cath(TM) 3.5F System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Best Vascular, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Best PMA Post-approval Study
Record Dates: First submitted 2009-02-24; First posted 2009-02-26 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Coronary In-stent Restenosis
Keywords: Coronary brachytherapy; Coronary restenosis; Coronary in stent restenosis
MeSH Terms: conditions — Coronary Restenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- On-label treatment: Patients treated in routine clinical practice following FDA Pre-Market Approval of the Beta-Cath(TM) 3.5F System within the parameters of the approved indications for use for the System ("on-label").

SUMMARY:
The study will evaluate the long-term safety and efficacy of intravascular beta radiation therapy to treat coronary in-stent restenosis using the Beta-Cath(TM) 3.5F System; data will be collected retrospectively on patients treated with the Beta-Cath™ 3.5F System in routine clinical practice following FDA pre-market approval of the System. Outcomes will be reported up to 5 years following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent on-label treatment (as defined below) with the Beta-Cath™ 3.5F System (30, 40 or 60mm) for in-stent restenosis (ISR) after coronary stenting.

  1. On-label treatment for the 30 and 40mm Beta-Cath™ 3.5F System is defined as: treatment of ISR in native coronary arteries with discrete lesions (treatable with a 20mm balloon) in reference vessel diameters (RVD) ranging from 2.7mm to 4.0mm
  2. On-label treatment for the 60mm Beta-Cath™ 3.5F System is defined as: treatment of ISR in native coronary arteries with lesions <40mm in length in RVD ranging from 2.7mm to 4.0mm
* Patients must have undergone brachytherapy treatment at least 6-8 months prior to enrollment in this retrospective study and the date of their treatment must be:

  1. On or after February 8, 2002 for the 30/40mm 3.5F System
  2. On or after June 25, 2003 for the 60mm 3.5F System

Exclusion Criteria:

* Patients who do not give informed consent
* Patients who do not meet the inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated on-label with the Beta-Cath™ 3.5F System at Washington Hospital Center
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-05; Primary Completion 2020-05 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | In-hospital and at 30 days, 6 months, 1, 2, 3, 4 and 5 years post-treatment
  Major Adverse Cardiac Events (MACE)

SECONDARY OUTCOMES:
Incidence of device-related procedural events | At time of intervention
  Incidence of device-related procedural events
Device success, including successful delivery of the Beta-Cath(TM) 3.5F System radiation source train, return of the radiation source train, and delivery of the intended dose | At time of intervention
  Device success, including successful delivery of the Beta-Cath(TM) 3.5F System radiation source train, return of the radiation source train, and delivery of the intended dose
Target Vessel Revascularization (TVR) | 6 months; 1, 2, 3, 4, and 5 years post-treatment
  Target Vessel Revascularization (TVR)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Washington Hospital Center / Cardiovascular Research Institute (CRI), Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided